CLINICAL TRIAL: NCT00410735
Title: Study of ONO-1078 in Patients With Chronic Sinusitis, a Double-blind, Randomized, Placebo-controlled, Parallel Group, Multi-center Study
Brief Title: Study of ONO-1078 in Patients With Chronic Sinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-1078-37
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Sinusitis
Keywords: ONO-1078; chronic sinusitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- P (Placebo Comparator)
  Interventions: Drug: Placebo
- E (Experimental)
  Interventions: Drug: Pranlukast hydrate

INTERVENTIONS:
Drug: Placebo — 0 mg BID for 12 weeks
  Arms: P
Drug: Pranlukast hydrate — 225 mg BID for 12 weeks
  Arms: E

SUMMARY:
To determine the efficacy and safety of ONO-1078 in patients with chronic sinusitis in a double-blind, randomized, placebo-controlled, parallel group, multi-center study

ELIGIBILITY:
Inclusion Criteria:

* chronic sinusitis

Exclusion Criteria:

* acute sinusitis
* chronic sinusitis with acute exacerbation

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
nasal congestion | 12 weeks
rhinorrhea | 12 weeks
postnasal drip | 12 weeks

SECONDARY OUTCOMES:
easiness of blowing nose | 12 weeks
easiness of removing postnasal drip | 12 weeks
dull headache | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hajime Yamamotoya, Study Director — Ono Pharmaceutical Co. Ltd
Locations (6):
- Japan (6):
  - Chubu region, Chūbu
  - Hokuriku region, Hokuriku
  - Kanto region, Kanto
  - Kinki region, Kinki
  - Kyushu region, Kyushu
  - Tohoku region, Tōhoku